CLINICAL TRIAL: NCT06593834
Title: A Clinical Study of Bacillus Coagulans in Acute Graft-Versus-Host Disease (aGVHD) After Hematopoietic Stem Cell Transplantation
Brief Title: A Clinical Study of Bacillus Coagulans in Acute Graft-Versus-Host Disease After Hematopoietic Stem Cell Transplantation
Acronym: aGVHD；BAT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yamin Fan (Other)
Responsible Party: Sponsor-Investigator, Yamin Fan, Principal Investigator, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Organization: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRS2400084534
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Acute Graft-versus-host Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): bacillus coagulans combined with the best treatment options for preventing aGVHD
  Interventions: Drug: bacillus coagulans combined with the best treatment options for preventing aGVHD
- Control group (Active Comparator): The best treatment options for preventing aGVHD
  Interventions: Drug: BAT

INTERVENTIONS:
Drug: bacillus coagulans combined with the best treatment options for preventing aGVHD — BAT means the best treatment options for preventing aGVHD
  Arms: Experimental group
Drug: BAT — BAT
  Arms: Control group

SUMMARY:
To evaluate the preventive effect of Bacillus coagulans on acute graft-versus-host disease (aGVHD) after hematopoietic stem cell transplantation

DETAILED DESCRIPTION:
The study is conducted on patients after hematopoietic stem cell transplantation and the intervention is Bacillus coagulans, aiming to investigate the preventive effect of Bacillus coagulans on acute graft-versus-host disease after hematopoietic stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are fully aware of the study, voluntarily participate and sign informed consent;
2. Age: ≥18 years old;
3. Patients with hematologic malignancies undergoing allo-HSCT and patients with severe aplastic anemia (SAA) undergoing allo-HSCT were treated with myeloablative conditioning (MAC).

Exclusion Criteria:

1. Refused to participate in this clinical study;
2. Unable to take the drug orally;
3. Allergic to Bacillus coagulans;
4. People take allo-HSCT with reduced intensity conditioning (RIC) and nonmyeloablative conditioning (NMC);lymphoma or multiple myeloma with auto-HSCT; multiple myeloma patients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Estimated)
Dates: Start 2024-09-27 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Rate of acute graft-versus-host disease | 100th day
  Will acute graft-versus-host disease occur within 100 days after hematopoietic stem cell transplantation and its probability of occurrence